CLINICAL TRIAL: NCT06980363
Title: Efficacy of Articaine Plus Hyaluronidase Enzymes Infiltration Versus Traditional Inferior Alveolar Nerve Block for the Extraction of Mandibular Molars
Brief Title: Hyaluronidase Enzymes and Local Anesthesia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2222
Record Dates: First submitted 2025-05-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Local Infiltration
MeSH Terms: interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional inferior alveolar nerve block by articaine (Active Comparator)
  Interventions: Drug: traditional inferior alveolar nerve block by articaine
- hyaluronidase plus articain buccal infiltration (Experimental)
  Interventions: Drug: hyaluronidase plus articain buccal infilteration

INTERVENTIONS:
Drug: traditional inferior alveolar nerve block by articaine — use articaine for inferior alveolar nerve block with buccal infiltration to anesthetized lower molar teeth
  Arms: traditional inferior alveolar nerve block by articaine
Drug: hyaluronidase plus articain buccal infilteration — use of articain plus hyaluronidase enzyme buccal infiltration to anesthetized lower molar teeth
  Arms: hyaluronidase plus articain buccal infiltration

SUMMARY:
* For both groups, local anaesthesia will be administered by one single surgeon and the extraction will be performed by another single surgeon across all subjects. The surgeon performing the extraction will be blinded with regard to the local anaesthesia technique used in this study
* A buccal infiltration injection of 1.5 ml of 4% articaine with 1:100,000 adrenaline (Septocaine, Septodont, New Castle, Del.) plus 1.5 ml of hyaluronidase enzyme (7.5IU/1ml) will be used in the study group while use 4% articaine with 1:100,000 adrenaline (Septocaine, Septodont, New Castle, Del.)only in traditional inferior alveolar nerve block in the control group
* In study and control groups, VAS (visual analogue scale=is an unmarked, continuous, horizontal,100-mm line, anchored by the end points of "no pain" on the left and "worst pain" on the right ) will be used to evaluate the pain levels of the patients associated with the injection and during extraction

ELIGIBILITY:
Inclusion Criteria:

* Medically stable patients
* Seeking for non surgical extraction of mandibular molar tooth

Exclusion Criteria:

* history of metabolic or systemic diseases affecting bone or healing process,

  * local infection
  * Grade III mobility
  * Neurological disorder
  * an analgesic use within 24 hours before anaesthesia administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-27 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale (VAS)0_10 | Periprocedural
  Ask the patient to scoring his pain during the extraction by visualanalogue scale0_10 as 0 no pain and 10 sever pain